CLINICAL TRIAL: NCT00718107
Title: Satisfaction Survey for ALS Patients Comparing Rooms With and Without Assistive Technology
Brief Title: Satisfaction Survey for Amyotrophic Lateral Sclerosis (ALS) Patients Comparing Rooms With and Without Assistive Technology
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to low enrollment. A survey has been implemented in place of a formal study.
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-15894
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders; Quality of Life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
The purpose of this study is :

1. To assess the ALS patient's satisfaction related to a hospital stay on the neurology floor of Hahnemann Hospital.
2. To compare the reported satisfaction of those individuals who stayed in a standard hospital room with those who stayed in Room 1455. Room 1455 is a room specifically set up with assistive technology related to environmental controls for individuals with disabilities.
3. To look at frequency of use of the various pieces of adaptive equipment.

ELIGIBILITY:
Inclusion Criteria:

* In-patients with probable or definite ALS, ages 18 - 90, staying on the neurology floor of Hahnemann Hospital

Exclusion Criteria:

* In-patients who do not meet the criteria of the diagnosis of ALS.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patients from the neurology floor of Hahnemann Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2005-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Period of Hospital Stay
  Survey administered asks patients to rate their satisfaction with their hospital stay from Very Dissatisfied to Very Satisfied. Specific questions included satisfaction with hospital staff, quality of care, and comfort and accessibility of their room.

CONTACTS AND LOCATIONS:
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States